CLINICAL TRIAL: NCT01457937
Title: Boceprevir/Peginterferon Alfa (PegIFN α)-2b/Ribavirin (Riba) in Difficult-to-Treat Menopausal Women With Chronic Hepatitis C Genotype 1 (Gt 1), Either Deemed Nonresponders to Peginterferon/Ribavirin or Treatment-naives (MEN_BOC)
Brief Title: Boceprevir/PegIFN α-2b/Riba in HCV+ Gt1 Menopausal Women, Nonresponders to PegIFN/Riba or Treatment-naives (MEN_BOC)
Acronym: MEN_BOC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Prof. Facchinetti Fabio, Prs admin, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2011-002459-33
Record Dates: First submitted 2011-10-08; First posted 2011-10-24 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Hepatitis C; Menopause
Keywords: HCV; Menopause; Peg IFN; Ribavirin; Boceprevir
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG IFN/Ribavirin (Active Comparator): Standard of care for HCV-positive CAH
  Interventions: Drug: Pegylated Interferon, Ribavirin, Boceprevir
- PEG IFN/Ribavirin/Boceprevir (Experimental): Combination to be tested for possible higher efficacy
  Interventions: Drug: Pegylated Interferon, Ribavirin, Boceprevir

INTERVENTIONS:
Drug: Pegylated Interferon, Ribavirin, Boceprevir — PEG IFN alfa 2b 1,5 ug/kg once weekly; Ribavirin (800-1400 mg / day)
  or
  PEG IFN alfa 2b 1,5 ug/kg once weekly; Ribavirin (800-1400 mg / day); Boceprevir (1.5 mcg / kg QW)
  Other Names: PEG IFN alfa 2b : Peg Intron; Ribavirin: Rebetol; Boceprevir: Victrelis

SUMMARY:
The cohort of post-menopausal women represents a group of very-difficult-to-treat patients in whom a more powerful approach is required in order to improve the disappointing response rate. Thus the addition, in patients with previous failure to PEG/RBV treatment or in naïve patients, of a powerful drug like Boceprevir could greatly improve SVR rate as suggested by the results of SPRINT_2 trial in whom Boceprevir addition determined a 30% improvement in SVR rate in difficult gt 1 patients of African descent versus standard PEG IFN/Ribavirin therapy or by those of RESPOND-2 that showed the same percent improvement of RGT-retreatment with Boc/P/R of previous failure of standard therapy.

Goal of the study is to verify whether the addition of a 24-week treatment with boceprevir to standard antiviral therapy with Peg IFN and ribavirin will increase the rate of SVR in patients difficult to treat, such as HCV-positive women in post-menopausal women with genotype 1, not only those who have never been treated, but also in those who have not responded to previous treatment with peginterferon and ribavirin (Riba).

DETAILED DESCRIPTION:
2.2.1 Hypothesis Our hypothesis is that the addition of a 24-week treatment with boceprevir to standard antiviral therapy with Peg IFN and ribavirin will increase the rate of sustained virological response (SVR) in patients difficult to treat, such as HCV-positive women in post-menopausal women with genotype 1, not only those who have never been treated, but also in those who have not responded to previous treatment with peginterferon and ribavirin (Riba) Objectives Retreatment Primary objective Verify whether the sustained virological response (SVR defined as HCV RNA undetectable at 24 weeks of follow-up) in menopausal women with HCV CAH genotype 1 who have not achieved a sustained virological response with a previous treatment with PEG IFN/ribavirin may increase by at least 20% after treatment with PEG IFN alfa 2b and boceprevir (1.5 mcg / kg QW) + Ribavirin (800-1400 mg / day) The primary efficacy endpoint, achieving SVR, will be evaluated with descriptive statistics (n,%) for each treatment arm.

Secondary objective It is represented by evaluation of the percent of patients with early virological response (undetectable HCV RNA at weeks 2, 4, 8 or 12) that reach SVR.

Naïve patients

Primary objective Verify whether SVR, defined as undetectable HCV-RNA at 24 weeks of follow-up may increase by at least 25% after treatment with PEG IFN alfa 2b plus ribavirin and boceprevir vs. PEG IFN alfa 2b plus ribavirin alone, in postmenopausal women with CHC genotype 1 not previously treated The primary efficacy endpoint, achieving SVR, will be evaluated with descriptive statistics (n,%) for each treatment arm.

Secondary objective It is represented by evaluation of the percent of patients with early virological response (undetectable HCV RNA at weeks 2, 4, 8 or 12) that reach SVR.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal females with previously documented CHC infection, either (A) relapser or with a >2log10 IU/ml HCV RNA decrease at week 12 in a previous PEG IFN/Ribavirin treatment or (B) naives;
* Subject must have a liver biopsy within the last 2 years with histology consistent with CHC and no other etiology.
* Subjects with bridging fibrosis or cirrhosis must have an ultrasound within 6 months of the Screening Visit (or between Screening and Day 1) with no findings suspicious for hepatocellular carcinoma (HCC).
* Subject must be willing to give written informed consent.

Exclusion Criteria:

* Coinfection with the human immunodeficiency virus (HIV) or hepatitis B virus (HBsAg positive).
* Treatment with any investigational drug within 30 days of the randomization visit in this study.
* Participation in any other clinical trial within 30 days of randomization or intention to participate in another clinical trial during participation in this study.
* Evidence of decompensated liver disease including, but not limited to, a history or presence of clinical ascites, bleeding varices, or hepatic encephalopathy.
* Diabetic and/or hypertensive subjects with clinically significant ocular examination findings: retinopathy, cotton wool spots, optic nerve disorder, retinal hemorrhage, or any other clinically significant abnormality.
* Pre-existing psychiatric condition(s).
* Clinical diagnosis of substance abuse of the specified drugs within the specified timeframes.
* Any known pre-existing medical condition that could interfere with the subject's participation in and completion of the study.
* Evidence of active or suspected malignancy, or a history of malignancy, within the last 5 years (except adequately treated carcinoma in situ and basal cell carcinoma of the skin). Subjects under evaluation for malignancy are not eligible.
* Subjects who had life-threatening serious adverse event (SAE) during screening period.
* Protocol-specified hematologic, biochemical, and serologic criteria: Hemoglobin <12 g/dL for females and <13 g/dL for males; Neutrophils <1500/mm^3 (blacks: <1200/mm^3); Platelets <100,000/mm^3; Direct bilirubin >1.5 x upper limit of normal (ULN)
* Serum albumin < lower limit of normal (LLN)
* Thyroid-stimulating hormone (TSH) >1.2 x ULN or <0.8 x LLN of laboratory, with certain exceptions.
* Serum creatinine >ULN of the laboratory reference.
* Protocol-specified serum glucose concentrations.
* Prothrombin time/partial thromboplastin time (PT/PTT) values >10% above laboratory reference range.
* Anti-nuclear antibodies (ANA) >1:320.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of sustained virological response in previous treatment failure or naive HCV-positive menopausal women. | Baseline and 72 weeks
  Verify whether the SVR (HCV RNA undetectable at 24 wks) in menopausal women with HCV CAH genotype 1 with a previous failure with PEG IFN/ribavirin or treatmenti-naive may increase by 20% or 25% respectively after treatment with PEG IFN alfa 2b and boceprevir (1.5 mcg / kg QW) + Ribavirin (800-1400 mg / day).

SECONDARY OUTCOMES:
Early virological response | Baseline and 12 weeks
  Evaluation of the percent of patients with early virological response (undetectable HCV RNA at weeks 2, 4, 8 or 12) that reach SVR

CONTACTS AND LOCATIONS:
Overall Officials: ERICA VILLA, Prof, Principal Investigator — Azienda Ospedaliero-Universitaria, University of Modena and Reggio Emilia
Locations (1):
- Gastroenterology Unit, Modena, Modena, Italy

REFERENCES:
- [Derived] Bernabucci V, Ciancio A, Petta S, Karampatou A, Turco L, Strona S, Critelli R, Todesca P, Cerami C, Sagnelli C, Rizzetto M, Camma C, Villa E. Boceprevir is highly effective in treatment-experienced hepatitis C virus-positive genotype-1 menopausal women. World J Gastroenterol. 2014 Nov 28;20(44):16726-33. doi: 10.3748/wjg.v20.i44.16726. PMID 25469044